CLINICAL TRIAL: NCT06736847
Title: Exploration of Lymph Node Metastasis and Tumor Deposit in the Posterior Gastric Mesentery Following D2 Lymphadenectomy Plus Complete Mesogastric Excision in Patients Who Received Distal Gastrectomy: A Prospective Observational Study
Brief Title: Exploration of Lymph Node Metastasis and Tumor Deposit in the Posterior Gastric Mesentery for Distal Gastric Cancer
Acronym: zydgc001
Status: Recruiting | Type: Observational
Sponsor: Jichao Qin (Other)
Responsible Party: Sponsor-Investigator, Jichao Qin, professor, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Other Study IDs: 2024-0899
Record Dates: First submitted 2024-09-01; First posted 2024-12-17 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Gastric Carcinoma
Keywords: Gastric cancer; Lymph node dissection; Posterior gastric mesentery; Lymph node metastasis
MeSH Terms: conditions — Stomach Neoplasms; Lymphatic Metastasis | interventions — Gastroenterostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Radical gastrectomy with membrane dissection
  Interventions: Procedure: distal gastrectomy with D2 lymphadenectomy plus complete mesogastric excision (CME) in gastric cancer

INTERVENTIONS:
Procedure: distal gastrectomy with D2 lymphadenectomy plus complete mesogastric excision (CME) in gastric cancer — distal gastrectomy with D2 lymphadenectomy plus complete mesogastric excision (CME) in gastric cancer

SUMMARY:
This study aims to evaluate lymph node metastasis and tumor deposit in the posterior gastric mesentery following distal gastrectomy with D2 lymphadenectomy plus complete mesogastric excision (CME) in gastric cancer.

DETAILED DESCRIPTION:
Since 1997, the AJCC has been using the number of lymph node metastases (pN staging) as a crucial indicator to assess the prognosis of gastric cancer patients. This system has been continuously updated, widely accepted by the global oncology community, and confirmed for its feasibility, applicability, convenience, and reproducibility. The number of metastatic lymph nodes in radical resection specimens of gastric cancer patients is the total count of lymph nodes with metastasis and is a key focus of postoperative pathological examination. D2 lymphadenectomy has become the standard operative procedure for advanced resectable gastric cancer and certain early-stage gastric cancers (diagnosed preoperatively with lymph node metastases). For advanced gastric cancer, there is growing evidence that the ideal surgical approach should involve D2 lymphadenectomy plus CME. In distal gastrectomy, the number of lymph nodes removed in D2 lymphadenectomy plus CME is significantly higher than in D2 dissection. Additionally, patients in the D2+CME group exhibit better long-term outcomes compared to the D2 group (DCGC01 study). Performing D2+CME surgery for distal gastric cancer involves the resection of the five major mesentery, including the posterior gastric mesentery, which may aid in thorough lymph node clearance and reduce cancer spillage. The posterior gastric mesentery comprises the No.11p and part of the No.11d lymph nodes. However, only the No.11p lymph nodes are resected in traditional D2 lymphadenectomy, resulting in incomplete lymph node clearance and postoperative tumor recurrence. Hence, the primary objective of this study is to examine lymph node metastasis in the posterior gastric mesentery following D2+CME in patients undergoing distal gastrectomy, aiming to offer evidence-based medical insights for standardizing surgical approaches in gastric cancer management.

ELIGIBILITY:
Inclusion Criteria:

1. Aged older than 18 years and younger than 85 years
2. Primary gastric adenocarcinoma confirmed by preoperative pathology result
3. cT2-4N0-3M0 at preoperative evaluation according to the American Joint 8 Committee on Cancer (AJCC) Cancer Staging Manual 7th Edition
4. Patients who received distal gastrectomy with D2 lymphadenectomy plus complete mesogastric excision
5. American Society of Anesthesiologists (ASA) class I, II, or III
6. Written informed consent

Exclusion Criteria:

1. Negative preoperative biopsy
2. Too late tumour stage or metastasis (cT4b/M1)
3. BMI>30 kg/m2
4. Total gastrectomy or proximal gastrectomy
5. previous neoadjuvant chemotherapy or radiotherapy
6. Previous upper abdominal surgery
7. Combined with other malignant diseases
8. Reject operation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who met the above inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of lymph node metastasis and tumor deposit in the posterior gastric mesentery | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastrointestinal Surgery, The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided